CLINICAL TRIAL: NCT00307255
Title: Phase I Trial of Abraxane in Combination With Gemcitabine in Patients With Solid Tumors
Brief Title: Paclitaxel Albumin-Stabilized Nanoparticle Formulation and Gemcitabine in Treating Patients With Advanced Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 0520; CDR0000550136 (Other: PDQ number)
Record Dates: First submitted 2006-03-24; First posted 2006-03-27 (Estimated); Last update posted 2012-04-04 (Estimated); Status verified 2012-04

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor; protocol specific; Paclitaxel; Abraxane; Gemcitabine; Gemzar; Phase I; Lineberger
MeSH Terms: interventions — Gemcitabine; Taxes; Albumin-Bound Paclitaxel

INTERVENTIONS:
Drug: gemcitabine hydrochloride — 1000 mg/m2 on days 1 and 8 of each 21 day cycle
  Other Names: Gemzar
Drug: paclitaxel albumin-stabilized nanoparticle formulation — 260 mg/m2 to 340 mg/m2 (dose will depend on when subject enters the study). Paclitaxel will be given on day 1 of each 21 day cycle (every 3 weeks)
  Other Names: Abraxane

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as paclitaxel albumin-stabilized nanoparticle formulation and gemcitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of paclitaxel albumin-stabilized nanoparticle formulation when given together with gemcitabine in treating patients with advanced metastatic solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the dose-limiting toxicity and maximum tolerated dose of paclitaxel albumin-stabilized nanoparticle formulation (Abraxane) in combination with gemcitabine hydrochloride in patients with advanced metastatic solid tumors.

Secondary

* Evaluate the efficacy of this regimen in these patients.

OUTLINE: This is a dose-escalation study of paclitaxel albumin-stabilized nanoparticle formulation (Abraxane).

Patients receive paclitaxel albumin-stabilized nanoparticle formulation (Abraxane) IV over 30 minutes on day 1 followed by gemcitabine hydrochloride IV over 30 minutes on days 1 and 8. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of paclitaxel albumin-stabilized nanoparticle formulation (Abraxane) until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Up to 10 additional patients may be treated at the MTD.

After completion of study treatment, patients are followed at 30 days.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed solid tumors

  * Advanced metastatic disease
* Measurable or evaluable disease
* Must meet 1 of the following criteria:

  * Failed prior standard therapy
  * Not a candidate for standard therapy
  * Has a disease for which there is no defined standard therapy
* No symptomatic brain metastases

PATIENT CHARACTERISTICS:

* ECOG functional status 0-2
* Life expectancy ≥ 8 weeks
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count > 100,000/mm^3
* Hemoglobin ≥ 9.0 g/dL
* Bilirubin normal
* Creatinine ≤ 1.5 times upper limit of normal (ULN) OR creatinine clearance ≥ 60 mL/min
* AST and ALT ≤ 2.5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* No prior anaphylactic reaction or severe allergic reaction to paclitaxel, docetaxel, or gemcitabine hydrochloride
* No active infectious process that will require treatment with antibiotics for > 4 weeks
* No uncontrolled congestive heart failure
* No symptomatic coronary artery disease or heart block
* No myocardial infarction within the past 3 months
* No peripheral neuropathy ≥ grade 2 from any cause

PRIOR CONCURRENT THERAPY:

* More than 3 weeks since prior chemotherapy, radiotherapy, or any other treatment
* No prior radiotherapy to > 25% of bone marrow
* No prior nitrosoureas
* No more than 6 prior courses of alkylating agents
* No more than 2 prior courses of mitomycin C
* No more than 3 prior courses of cytotoxic therapy for metastatic disease
* No concurrent filgrastim (G-CSF), pegfilgrastim, or sargramostim (GM-CSF) during study course 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2006-08; Primary Completion 2007-09 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | 21 days
  Toxicity will be graded using the CTCAE version 3.0 and will be assessed on cycle one (21 days)
Maximum Tolerated Dose(MTD) | 1 year
  If greater than or equal to 2 of 6 patients (33%) experience a DLT, then that dose level will be considered to have excessive toxicity and will = MTD

SECONDARY OUTCOMES:
Radiographic Response to Treatment | every 42 days
  Radiographic response will be measured and evaluated using RECIST criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E. Stinchcombe, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- University of North Carolina Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States